CLINICAL TRIAL: NCT02748408
Title: The Medacta SMS Femoral Stem Component. A Multi-National, Multi-Centre, Clinical Surveillance Study
Brief Title: The Medacta International SMS Post-Marketing Surveillance Study
Status: Recruiting | Type: Observational
Sponsor: Medacta International SA (Industry)
Responsible Party: Sponsor
Other Study IDs: P01.019.01
Record Dates: First submitted 2016-04-11; First posted 2016-04-22 (Estimated); Last update posted 2025-09-29 (Actual); Status verified 2025-03

CONDITIONS: Arthrosis; Traumatic Arthritis; Rheumatoid Polyarthritis; Congenital Hip Dysplasia; Avascular Necrosis of the Femoral Head
MeSH Terms: conditions — Osteoarthritis; Hip Dislocation, Congenital; Femur Head Necrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

INTERVENTIONS:
Device: SMS femoral stem

SUMMARY:
This is a Post-Marketing Surveillance of SMS femoral stem prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a severely painful and/or disabling hip joint with osteoarthritis, traumatic arthritis or developmental dysplasia of the hip or avascular necrosis of the femoral head.
* In order to take part in this study, all study participants must be between the ages of 18 and 75 years of age, at the time of surgery.
* Scheduled for a primary total hip replacement.

Exclusion Criteria:

* Active infection
* Pregnancy
* Mental illness where the known condition is likely to compromise the patient's ability to consent, affect the patient's assessment of their progress or complete the 10 year cycle of follow-up appointments and reviews
* Grossly distorted anatomy (surgeon's discretion)
* Osteomalacia where uncemented implant fixation is contraindicated
* Active rheumatoid arthritis.
* Osteoporosis
* Metabolic disorders which may impair bone formation where uncemented implant fixation is contraindicated
* Muscular atrophy or neuromuscular disease
* Allergy to implant material
* Any patient who cannot or will not provide informed consent for participation in the study
* Those whose prospects for a recovery to independent mobility would be compromised by known coexistent, medical problems

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals suitable for hip replacement using the Medacta SMS femoral stem
Sampling Method: Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2015-07; Primary Completion 2032-07 (Estimated); Study Completion 2032-07 (Estimated)

PRIMARY OUTCOMES:
survivorship of the Medacta SMS femoral stem | 10-year

SECONDARY OUTCOMES:
clinical performance | 3, 5, 7 and 10 years
  Harris Hip Score
radiographic performance | 3, 5, 7 and 10 years
  presence of radiolucencies
Evaluate the patient satisfaction | 6 months, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10 years
  Oxford score
Evaluate the quality of life | 6 months, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10 years
  EQ-5D
pattern of bone remodeling | 6 weeks, 6 months, 1 year
  Dual Energy X ray Absorptiometry (DEXA)
stem migration | 6 weeks, 6 months, 1 and 2 years
  Radiostereometric Analysis (RSA)
Adverse events | up to 10 years
  record of adverse event

CONTACTS AND LOCATIONS:
Locations (4):
- Herz-Jesu Krankenhaus, Vienna, Austria
- Istituto Ortopedico Galezzi, Milan, Milan, Italy
- Bürgerspital Solothurn, Solothurn, Switzerland
- The Elective Orthopaedic Centre (EOC), Epsom, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No